CLINICAL TRIAL: NCT00115856
Title: Imaging of Plaque in Atherosclerosis With Intravascular MRI
Brief Title: Imaging of Plaque With Magnetic Resonance Imaging (MRI)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Peter Ganz MD (Unknown)
Responsible Party: Principal Investigator, Andrew Peter Selwyn, MD, MD, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2001P-000114
Record Dates: First submitted 2005-06-26; First posted 2005-06-27 (Estimated); Last update posted 2015-08-03 (Estimated); Status verified 2015-07

CONDITIONS: Arterial Occlusive Disease
Keywords: Arterial Disease
MeSH Terms: conditions — Arterial Occlusive Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Subjects studied (No Intervention): Single arm exploratory feasibility safety and efficacy study of MRI to image atherosclerosis in arteries
  Interventions: Procedure: Intravascular MRI

INTERVENTIONS:
Procedure: Intravascular MRI — Arterial imaging of atherosclerosis

SUMMARY:
This study aims to develop and refine the use of an intravascular wire to image plaque in the aorta, iliac and femoral artery using MRI. This project aims to use this increased resolution to identify the features within the plaque that is known to be associated with increased risk of plaque and vessel occlusion.

The hypothesis is Intravascular MRI can detect and measure changes in response to therapy over time in the critical features in plaques in peripheral arteries of patients with atherosclerosis.

DETAILED DESCRIPTION:
For those patients undergoing cardiac catheterization, an 8French sheath will be introduced via a femoral artery approach. This size sheath allows us to visualize the distal aorta while performing the intra vascular ultrasound ( IVUS). For these patients, if a femoral venous sheath is also positioned for clinical purposes, then this access will also be utilized to introduce the MRI coil. This imaging approach will allow us to compare the feasibility of intravascular MRI imaging from: a) the artery; b) the vein; c) a combination of both.

For those patients not scheduled to undergo a clinically indicated cardiac catheterization, only a 6French sheath will be introduced via a femoral artery approach. In these patients, no femoral venous sheath will be introduced and the arterial access will not be upsized to a 8French sheath.

Two tablespoons of blood will be drawn from each patient to assess inflammatory markers such as C-Reactive Protein (CRP) as well as to confirm a negative pregnancy test for female patients of childbearing age.

Using 20cc of non-ionic contrast, an angiogram of the distal aorta and the ilio-femoral region will be performed and recorded on disc (5mins). Thereafter, an approved guidewire and intravascular ultrasound catheter will be positioned in the same arteries via the same access route, and ultrasound images of the arterial segment will be recorded (10mins.). The guidewire and the ultrasound coil will then be removed. Finally, an intravascular MRI wire will be advanced through the same arterial access and/or the previously indicated venous access under X-ray control and positioned in the desired atherosclerotic segment in the region of the distal aorta or at the ilio-femoral area. The MRI wire(s) will be secured in place by Tegaderm and the femoral sheath(s) will be sutured in stable position. The patient will then be transported to the MRI scanner, positioned in the scanner and images recorded over a period not exceeding 60 minutes. During the transport and throughout the MRI scanning, the patient will be monitored via an MRI-compatible cardiac monitor. During the time that the intravascular MRI coil is within the femoral sheath, it will be continuously perfused with heparinized saline and the patient will receive weight- adjusted (12 U/kg) intravenous heparin for systemic anticoagulation to prevent thrombosis. To obtain the MRI images, the patients will receive gadolinium contrast as per routine radiology protocols (0.1-0.2 mmol/kg). After recording the MRI images, the MRI coil(s) and the femoral sheath(s) will be removed from the artery and/or the vein as per usual care.

ELIGIBILITY:
Inclusion Criteria:

* Male and female adults (aged 25-80) seen at the Brigham and Women's Hospital (BWH) clinic who have known arterial disease who consent to cannulation of the femoral artery for this research.
* Patients in the prespecified age group who are scheduled to undergo a clinically indicated heart or peripheral catheterization at the BWH catheterization (cath) lab who will have a tube (sheath) already positioned in their femoral artery
* Patient must be in stable condition with regard to symptoms, vital signs and the monitored electrocardiogram

Exclusion Criteria:

* Unstable symptoms, vital signs or electrocardiogram after the heart cath
* Any complications during the heart cath (eg., bleeding, angina, arrhythmias, technical difficulties cannulating the femoral artery)
* Creatinine >2.0mg/dl
* Pregnancy
* Contraindications to anticoagulation
* Patients with a metal implant, pacemaker, cardiac defibrillator, metal fragments in the eye, bullets/metal objects in the body

Ages: 25 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2001-01; Primary Completion 2005-06 (Actual); Study Completion 2005-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Selwyn, MD, Principal Investigator — Brigham and Womens Hospital
Locations (1):
- Brigham and Womens Hospital, Boston, Massachusetts, United States